CLINICAL TRIAL: NCT04233632
Title: Randomized Comparative Study of the Contraceptive Efficacy of the Cupid, Cupid 2 and FC2 Female Condom
Brief Title: Comparative Study of the Contraceptive Efficacy of the Cupid, Cupid 2 and FC2 Female Condom
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Prof Mags Beksinska (Other)
Responsible Party: Sponsor-Investigator, Prof Mags Beksinska, Deputy Executive Director, University of Witwatersrand, South Africa
Organization: University of Witwatersrand, South Africa (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CoCo
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Pregnancy Prevention
Keywords: Female condom; Pregnancy Prevention; Sexually transmitted infection prevention; Condom acceptability; FC2; Cupid

STUDY DESIGN:
Intervention Model Description: This research study will be a parallel randomized controlled trial to assess the effectiveness of three female condoms (Cupid, Cupid 2 and FC2) for the prevention of pregnancy among women choosing the female condom as their method of fertility regulation
Who Masked: Outcomes Assessor
Masking Description: The three condoms in the trial are distinctly different and so condom specific training is required and so cannot be blinded. The statistician analysing the data will be blinded to female condom type.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- FC2 Condom (Active Comparator): Participants will be randomized to either of the 3 groups and provided with their randomized method at enrolment and at each follow up visit until the final visit.
  Interventions: Device: FC2 Condom
- Cupid Condom (Active Comparator): Participants will be randomized to either of the 3 groups and provided with their randomized method at enrolment and at each follow up visit until the final visit
  Interventions: Device: Cupid Condom
- Cupid 2 Condom (Active Comparator): Participants will be randomized to either of the 3 groups and provided with their randomized method at enrolment and at each follow up visit until the final visit
  Interventions: Device: Cupid 2 Condom

INTERVENTIONS:
Device: FC2 Condom — FC2: FC2 is composed of a synthetic nitrile rubber latex and 170mm in length. It has a flexible inner ring as the internal retention mechanism and a circular ring as the outer retention mechanism at the open end of the condom. It is pre-lubricated with silicone oil. It has a shelf-life of 5 years and is available in clear and other colors/scents. It is manufactured by Female Health Company, USA and has USFDA, World Health Organisation (WHO)/United Nations Populations Fund (UNFPA) and South African Bureau of Standards (SABS) approval
  Arms: FC2 Condom
Device: Cupid Condom — Cupid is composed of a Natural rubber latex and is 155mm in length. It has a Medical grade sponge as the internal retention mechanism and an octagonal outer frame as the outer retention mechanism. It is pre-lubricated with silicone oil. It has a shelf-life of 3 years and is available in clear and red color, vanilla scented variety. It is manufactured by Cupid Ltd, India and has WHO)/UNFPA, India Drug Control Authority, Conformitè Europëenne (CE) Mark of the European Union (EU) and SABS approval
  Arms: Cupid Condom
Device: Cupid 2 Condom — Cupid2 is composed of a Natural rubber latex and is 125mm in length. It has a Medical grade sponge as the internal retention mechanism and an octagonal outer frame as the outer retention mechanism. It is pre-lubricated with silicone oil. It has a shelf-life of 3 years and is available in Clear and purple color, vanilla scented variety. It is manufactured by Cupid Ltd, India and has WHO)/UNFPA, India Drug Control Authority, CE Mark of the EU and SABS approval
  Arms: Cupid 2 Condom

SUMMARY:
This research study aims to assess the effectiveness of three female condoms [Cupid, Cupid 2 and Female Condom 2(FC2)] for the prevention of pregnancy among women choosing the female condom (FC) as their method of fertility regulation. Participants will be followed-up monthly for up to seven months. A daily diary will be used to record menstrual pattern, acts of intercourse and details of condom usage.

DETAILED DESCRIPTION:
This research study aims to assess the effectiveness of three female condoms (Cupid, Cupid 2 and FC2) for the prevention of pregnancy among women choosing the female condom (FC) as their method of fertility regulation.

The study is a randomized comparative prospective follow-up study. Participants will be followed-up monthly for up to seven months. A daily diary will be used to record menstrual pattern, acts of intercourse and details of condom usage. The primary endpoint will be the occurrence of pregnancy or use of emergency contraception, and the diary information will allow pregnancy rates to be characterized by patterns of condom use and failures (contraceptive efficacy and effectiveness rates).

The target population will be 780 urban and peri urban, sexually active women who are experienced users of FCs. Recruitment will be from a family planning clinic associated with the MatCH Research Unit (MRU), University of the Witwatersrand, Durban, South Africa and the surrounding community. The woman rather than the couple will be the unit of observation since the major outcome to be measured is pregnancy. There will be monthly follow-ups of participants from enrollment until after the 6th menstrual cycle (month 1,2,3,4,5 and 6). All visits will be conducted at the research site. The diary, to be completed on a daily basis by the participants, will indicate whether the coital frequency differs significantly between subgroups (students, urban, peri-urban).

Female clients of the Commercial City Clinic and other women presenting at the site will be informed about the study. If a potential participant expresses interest in participating, she will be given the study information sheet to read, which will describe the study requirements and her potential role in the study. If she agrees to take part in the research, she will be asked to provide written informed consent. The participant will be administered the screening form to determine whether she meets study inclusion criteria.

Eligible women who agree to participate will undergo a baseline interview. Information collected during the enrollment interview will include demographic data and information on the participant's general and reproductive health. The data collected on reproductive health variables will include the date of last menstrual period (LMP), history of pregnancies, births and miscarriages, a contraceptive history as well as a sexual history. After completion of the interview, the participant will be randomized to the use on one FC type.

Male partners will not be asked to sign an Informed Consent as they will not be required to participate in the research, but female participants will be given an additional information sheet if they desire to give to the male partner to tell them about the study.

If a potential participant does not wish to be enrolled, she will be provided with referral (should she wish) for any reproductive health services according to normal clinical practice at the study site. Her reasons will be recorded on the log of refusals. This information will be used to compile statistics on the participation rates and reasons for nonparticipation.

Although all study participants are required to have ever used a FC, some may have not used the FC they have been randomized to and have experience with other FC types. All participants will be retrained regardless of previous FC use using a pelvic model. The study staff will demonstrate FC insertion and train the participants in the proper use of the randomized FC type. Further, they will provide instruction on how to complete the condom use log and the study diary. She will also receive instructions on use in her preferred language (English or Zulu).

The participants will be given their first study packet which will contain either Cupid, Cupid 2 or FC2 with a diary for the first month of the study. Research staff will discuss with the participant how many condoms they require for the month. The participants will be instructed how to complete the diary card. The first follow-up visit should occur approximately one month after enrollment and should be pre-scheduled. The date of the first follow-up visit should be written in an appointment card and on the designated location on the Condom diary card. Participants who finish using their condoms prior to their scheduled follow-up visit, will be encouraged to contact MRU for a resupply.

There will be six follow-up visits in person at 1, 2, 3, 4, 5, and 6 months. Telephonic follow-up will be conducted between 7-14 days post enrollment to confirm any queries or problems in use of condoms or diaries.

Participants will be administered a follow-up survey about their experiences using their randomized FC, whether there has been a delay in expected onset of menses, the date of last menstrual period, and information on the use of other contraceptives since the last visit. The daily diary will also be reviewed at each visit for completeness and accuracy. A pregnancy test will be carried out at every on-site visit. Any reported or confirmed pregnancies will include counseling and referral to an antenatal or other healthcare facility. The final follow up visit will be scheduled after 6th menstrual cycle.

Women will be discontinued from the study at any stage during follow-up for: pregnancy, unwillingness to continue use of FCs or change to a non-study contraceptive method as her main contraceptive method, or refusal to be followed up.

Block randomization will be used. A statistician (not otherwise involved in this study) will develop the random allocation sequence using a validated statistical program in Stata (StataCorp LP, College Station, Texas, USA). Use-order assignments will be generated via the RedCap electronic program. The statistician will be blinded until all data have been captured and the primary analysis programs have been verified. Due to dissimilarities of the study products, it will not be possible to blind participants and clinic staff associated with the project.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy sexually active women who have ever used an FC and using condoms (male or female) as their current method of contraception.
2. Be 18 to 40 years at enrolment (inclusive).
3. Have a negative urine pregnancy test at enrolment visit.
4. Is HIV negative
5. Have a history of regular cyclic menses (usual length of 21 to 35 days) when not using hormonal contraception.
6. Have at least one spontaneous menstrual cycle (two menses) following a pregnancy that ended at 14 or more weeks gestation.
7. Have at least one cycle (two menses) after an abortion at less than 14 weeks gestation.
8. Be willing to accept a risk of pregnancy.
9. Reporting to have at least four acts of heterosexual vaginal intercourse per month for a period of 6 months.
10. Be willing to only use the study product (Cupid or FC2 female condom) as the primary method of contraception over the course of the study.
11. Be capable of using the study product properly and agree to observe all study directions and requirements.
12. Be willing to keep a daily diary to record menstrual pattern, acts of intercourse, and details of condom use and any condom failures.
13. Be willing to state that, to her best knowledge, her sexual partner:

    * Has not had a vasectomy or been previously diagnosed as infertile.
    * Is HIV negative
    * Has no known history of allergy or sensitivity to natural rubber latex, water-based or silicone lubricants
    * Does not want her to become pregnant in the next 7 months
14. Agree to have fingerprint identity check
15. Be willing to give written informed consent to participate in the trial.
16. Intend to stay in the area for the next 6-7 months
17. Be willing to be randomized

Exclusion Criteria:

1. Have a history of allergy or sensitivity to rubber latex or water-based /silicone lubricants
2. Have evidence of sexually transmitted infections on syndromic assessment and / or vaginal examination
3. Be pregnant, have a suspected pregnancy or desire to become pregnant during the course of the study.
4. Have a history of infertility or pelvic inflammatory disease without a subsequent spontaneous intrauterine pregnancy.
5. Have been diagnosed with pelvic inflammatory disease (PID) without a subsequent intrauterine pregnancy.
6. Be in a monogamous relationship of less than 4 months with their partner.
7. Have any contraindications to pregnancy (medical condition) or regularly use medications that are unsafe to use in pregnancy
8. Have shared injection drug needles in the past unless has a negative HIV test at least 6 weeks since last use.
9. HIV positive.
10. Have been diagnosed with genital herpes simplex virus (HSV), with the first occurrence (initial episode) within 3 months prior to screening or have clinical evidence of HSV on exam.
11. Be lactating or breastfeeding.
12. Have any clinically significant abnormal vaginal bleeding or spotting within the month prior to screening.
13. Have had vaginal or cervical biopsy or vaginal surgery within 3 months prior to screening.
14. Have used vaginal or systemic antibiotics or antifungal agents within 14 days prior to screening or enrollment.
15. Have received a Depo-Provera® injection in the 6 months prior to enrolment or Nur-Isterate in the last 4 months prior to enrolment
16. Have a past (within 12 months) or current history of alcohol or drug [recreational, prescription or over-the-counter (OTC)] abuse.
17. Have taken an investigational drug or used an investigational device within the past 30 days.
18. Have issues or concerns (in the judgment of the investigator) that may compromise the safety of the subject or confound the reliability of compliance and information acquired in this study.

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Participants must be female as female condoms inserted vaginally are being evaluated
Enrollment: 400 (Actual)
Dates: Start 2019-11-27 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2021-11-10 (Actual)

PRIMARY OUTCOMES:
Pregnancy | 6-7 months
  The main outcome measure of the study is the occurrence of pregnancy, which will be used to estimate the overall effectiveness of the method. For the overall pregnancy rate all pregnancies will be counted regardless of the reason(s) for the failure. Pregnancy rates will be computed using life table techniques. If the pregnancy rates are reasonably constant with time, then the Pearl index (pregnancies per 100 years of use) will be used and confidence intervals estimated from the Poisson distribution. Discrete time life-table methods will be used to explore patterns of failures associated with correct, incorrect and non-use of condoms (in each interval subjects will be classified according to the type or pattern of condom use and the life-table or Pearl rates computed for each stratum). Failure modes associated with the use of the female condoms per act of intercourse in which a FC was used.

SECONDARY OUTCOMES:
Clinical breakage | 6-7 months
  Clinical breakage is defined as breakage during sexual intercourse or during withdrawal of the female condom from the vagina. Clinical breakage is breakage with potential adverse clinical consequences. The clinical breakage rate is calculated by dividing the number of female condoms reported to have broken during sexual intercourse or during withdrawal by the number of female condoms used during sexual intercourse.
Non-clinical breakage | 6-7 months
  Non-clinical breakage is breakage noticed before intercourse or occurring after withdrawal of the condom from the vagina (no potential adverse clinical consequences).
Total breakage | 6-7 months
  Total breakage is defined as the sum of all female condom breakages at any time before, during or after sexual intercourse. It includes both clinical breakages and non-clinical breakages. The total breakage rate is calculated by dividing the total number of female condoms that broke by the number of female condom packages opened.
Slippage | 6-7 months
  Slippage is defined as an instance when a female condom that slips completely out of the vagina during sexual intercourse. The slippage rate is calculated by dividing the number of female condoms that slipped by the number of female condoms used during sexual intercourse.
Misdirection | 6-7 months
  Misdirection is defined as vaginal penetration whereby the penis is inserted between the female condom and the vaginal wall. The misdirection rate is calculated by dividing the number of reported events of misdirection by the number of female condoms used during sexual intercourse.
Invagination | 6-7 months
  Invagination is defined as an instance when the external retention feature of the female condom is partially or fully pushed into the vagina during sexual intercourse. The invagination rate is calculated by dividing the number of events of invagination by the number of female condoms used during sexual intercourse.
Total clinical failure | 6-7 months
  Total clinical failure is defined as the sum of female condoms that clinically break or slip, or are associated with misdirection, invagination or any additional failure modes(s) identified in the risk assessment which results in the reduction of the female condom protective function. The total clinical failure rate is calculated by dividing the number of female condoms with a clinical failure by the number of female condoms used during sexual intercourse.
Total female condom failure | 6-7 months
  Total female condom failure is defined as a female condom for which a non-clinical breakage, clinical breakage or slippage occurs, or is associated with misdirection, invagination or any additional failure modes(s) identified in the risk assessment. The female condom failure rate is calculated by dividing the number of female condoms that fail by the number of female condom packages opened.

CONTACTS AND LOCATIONS:
Overall Officials: Mags E Beksinska, PhD, Principal Investigator — MatCH Research Unit
Locations (1):
- MatCH Research Unit [Maternal, Adolescent and Child Health Research Unit], Durban, KwaZulu-Natal, South Africa

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Warren M. Condoms: the multipurpose prevention technologies that already exist. BJOG. 2014 Oct;121(Suppl 5):9-11. doi: 10.1111/1471-0528.12913. No abstract available. PMID 25335833
- [Background] Peters A, Jansen W, van Driel F. The female condom: the international denial of a strong potential. Reprod Health Matters. 2010 May;18(35):119-28. doi: 10.1016/S0968-8080(10)35499-1. PMID 20541090
- [Background] Reproductive Health Supplies Coalition. Caucus on new and underused reproductive health technologies. Product brief: female condom. Reproductive Health Supplies Coalition; 2013. [Online]. [Cited: 19th Dec 2016]. URL: https://www.rhsupplies.org/fileadmin/uploads/rhsc/Working_Groups/New_Underused_RH_Technologies_Caucus/Documents/Technical_Briefs/rhsc-brief-female-condom_A4.pdf
- [Background] United Nations Population Fund. HIV prevention gains momentum. New York: UNFPA, 2011. 978-0-89714-933-4.
- [Background] Center for Health and Gender Equity. Female condoms and US foreign assistance: an unfinished imperative for women's health. Washington, DC; 2011. https://www.unfpaprocurement.org/documents/10157/37547/UNFPA+Female+Cond om+Prequalification+List/05feba45-4893-474a-81d4-7b61e4f68ae7
- [Background] Beksinska M, Smit J, Joanis C, Potter W. New female condoms in the pipeline. Reprod Health Matters. 2012 Dec;20(40):188-96. doi: 10.1016/S0968-8080(12)40659-0. PMID 23245425
- [Background] Mqhayi M,Beksinska M,Smit J,Mqoqi N,Tshukudu D,NutleyT,Hatzell T,Wesson J,Marumo E.Introduction of the female condom in SA: Programmeme activities and performances 1998-2000.Durban: RHRU,FHI,NDoh,2003
- [Background] Mantell JE, Scheepers E, Karim QA. Introducing the female condom through the public health sector: experiences from South Africa. AIDS Care. 2000 Oct;12(5):589-601. doi: 10.1080/095401200750003770. PMID 11218545
- [Background] Farr G, Gabelnick H, Sturgen K, Dorflinger L. Contraceptive efficacy and acceptability of the female condom. Am J Public Health. 1994 Dec;84(12):1960-4. doi: 10.2105/ajph.84.12.1960. PMID 7998637
- [Background] Bounds W, Guillebaud J, Newman G B. Female Condom (Femidom). A clinical study of its use-effectiveness and patient acceptability. The British Journal of Family Planning 1992; 18:3641.
- [Background] Trussel J. Contraceptive efficacy of the Reality female condom. Contraception 1998;58: 148.
- [Background] Trussell J, Sturgen K, Strickler J, Dominik R. Comparative contraceptive efficacy of the female condom and other barrier methods. Fam Plann Perspect. 1994 Mar-Apr;26(2):66-72. PMID 8033980
- [Background] Steiner M, Trussell J, Glover L, Joanis C, Spruyt A, Dorflinger L. Standardized protocols for condom breakage and slippage trials: a proposal. Am J Public Health. 1994 Dec;84(12):1897-900. doi: 10.2105/ajph.84.12.1897. PMID 7998626
- [Background] Beksinska M, Joanis C, Manning J, Smit J, Callahan M, Deperthes B, Usher-Patel M. Standardized definitions of failure modes for female condoms. Contraception. 2007 Apr;75(4):251-5. doi: 10.1016/j.contraception.2006.10.003. Epub 2007 Feb 7. PMID 17362701
- [Background] Frezieres RG, Walsh TL, Nelson AL, Clark VA, Coulson AH. Evaluation of the efficacy of a polyurethane condom: results from a randomized, controlled clinical trial. Fam Plann Perspect. 1999 Mar-Apr;31(2):81-7. PMID 10224546
- [Background] Beksinska M, Nkosi P, Mabude Z, Smit J, Zulu B, Phungula L, Greener R, Kubeka M, Milford C, Lazarus N, Jali Z, Mantell JE. Twenty years of the female condom programmeme in SA: past, present and future. SAn Health Review, 2017. Chapter 14. In: Padarath A, Barron P, editors. SAn Health Review 2017. Durban: Health Systems Trust; 2017. URL: http://www.hst.org.za/publications/south-african-health-review-2017. Pg 147
- [Background] Beksinska ME, Piaggio G, Smit JA, Wu J, Zhang Y, Pienaar J, Greener R, Zhou Y, Joanis C. Performance and safety of the second-generation female condom (FC2) versus the Woman's, the VA worn-of-women, and the Cupid female condoms: a randomised controlled non-inferiority crossover trial. Lancet Glob Health. 2013 Sep;1(3):e146-52. doi: 10.1016/S2214-109X(13)70054-8. Epub 2013 Aug 23. PMID 25104263
- [Background] Joanis C, Beksinska M, Hart C, Tweedy K, Linda J, Smit J. Three new female condoms: which do South-African women prefer? Contraception. 2011 Mar;83(3):248-54. doi: 10.1016/j.contraception.2010.08.002. Epub 2010 Sep 17. PMID 21310287
- [Background] Beksinska M, Greener R, Kleinschmidt I, Pillay L, Maphumulo V, Smit J. A randomized noninferiority crossover controlled trial of the functional performance and safety of new female condoms: an evaluation of the Velvet, Cupid2, and FC2. Contraception. 2015 Sep;92(3):261-7. doi: 10.1016/j.contraception.2015.05.008. Epub 2015 May 20. PMID 26002805
- [Background] Farley TM. Life-table methods for contraceptive research. Stat Med. 1986 Sep-Oct;5(5):475-89. doi: 10.1002/sim.4780050512. PMID 3538263